CLINICAL TRIAL: NCT01551914
Title: Medico-economic Evaluation Comparing the Use of Ultrasonic Scissors to the Conventional Techniques of Haemostasis in Thyroid Surgery by Cervicotomy
Acronym: FOThyr
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RC11_0148
Record Dates: First submitted 2012-02-23; First posted 2012-03-13 (Estimated); Last update posted 2014-07-01 (Estimated); Status verified 2014-06

CONDITIONS: Thyroid Tumor
Keywords: Ultrasonic scissors; thyroidectomy
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- ultrasonic scissors (Experimental)
  Interventions: Device: Ultrasonic Scissors (Ethicon)
- conventional techniques of haemostasis (Active Comparator): clips, ligatures, and bipolar coagulation
  Interventions: Device: Bipolar Electrosurgical instruments (Medtronic) (SLS- Clips)

INTERVENTIONS:
Device: Ultrasonic Scissors (Ethicon) — Haemostasis using Ultrasonic scissors
  Other Names: Harmonic Focus scissors (Ethicon)
  Arms: ultrasonic scissors
Device: Bipolar Electrosurgical instruments (Medtronic) (SLS- Clips) — bipolar, monopolar or clip coagulation techniques
  Other Names: Bipolar Electrosurgical instruments (Medtronic); SLS- Clips
  Arms: conventional techniques of haemostasis

SUMMARY:
The aim of our study is to evaluate the ultrasonic scissors (Harmonic Focus Ethicon Endo-Surgery Laboratory) as a device of hemostasis in thyroid surgery (total thyroidectomy) by cervicotomy, and to show a decrease in transient hypoparathyroidism compared to conventional techniques of haemostasis (clips, ligatures, and bipolar coagulation). Secondary objectives of the study are the evaluation of (i) recurrent nerve morbidity, (ii) postoperative bleeding, (iii) postoperative pain, (iv) cost of both techniques (microcosting), (v) the overall cost of the techniques at six months, (vi) a linking of costs and medical outcomes and (vii) an estimation of the potential impact of new technology on the organization of operating rooms (operating time).

ELIGIBILITY:
Inclusion Criteria:

* Age > or = 18 yrs
* With a toxic goiter or not, Graves' disease or thyroid nodule requiring a total thyroidectomy
* Thyroidectomy under cervicotomy
* No echographic criteria to suspect a cancer: poorly defined nodules, microcalcifications, cervical nodes
* Patient covered by social security
* Patient's informed and written consent
* Possible follow-up during 6 months

Exclusion Criteria:

* Minors and adults under guardianship
* Preoperatively known thyroid cancer by cytology
* Planned partial thyroidectomy
* Peri-operatively antiplatelet intake
* Preoperatively ENT examination (if performed) finding a vocal cords affection
* Diving goiter (> 3 cm below the sternal notch)
* Surgery using videoscopy
* Lack of possible monitoring during the 6 months after surgery
* History of anterior cervical surgery
* Pregnancy and breast-feeding
* hypercalcemia (calcemia> 2.6 mmol/l)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1350 (Estimated)
Dates: Start 2012-03; Primary Completion 2014-10 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Immediate hypoparathyroidism (serum calcium <2 mmol/L at day 2) | Day 2

SECONDARY OUTCOMES:
Medico-economic evaluation | Day 0 (Procedure)
  Operating time
Medico-economic evaluation | Day 0 (procedure)
  Cost of the two techniques by microcosting
Medico-economic evaluation | Month 6
  Total cost at month 6
Medico-economic evaluation | From Day 0 until Month 6
  Incremental cost effectiveness ratio
Operative morbidity | Month 6
  Final hypoparathyroidism: calcium in the sixth postoperative month inferior than 2 mmol / L
Operative morbidity | Until Month 6
  Recurrent disease
Operative morbidity | Day 0 to Day 2
  Hemorrhagic disease

CONTACTS AND LOCATIONS:
Overall Officials: Eric Mirallié, Professor, Principal Investigator — Nantes University Hospital
Locations (1):
- CHU Nantes, Nantes, Nantes, France

REFERENCES:
- [Derived] Christou N, Blanchard C, Pattou F, Volteau C, Brunaud L, Hamy A, Dahan M, Prades JM, Landecy G, Dernis HP, Lifante JC, Sebag F, Jegoux F, Babin E, Bizon A, Caillard C, Mathonnet M, Mirallie E. Advanced age does not increase morbidity after total thyroidectomy. Result of a prospective study. Am J Surg. 2019 Apr;217(4):767-771. doi: 10.1016/j.amjsurg.2018.07.029. Epub 2018 Jul 25. PMID 30055804
- [Derived] Blanchard C, Pattou F, Brunaud L, Hamy A, Dahan M, Mathonnet M, Volteau C, Caillard C, Durand-Zaleski I, Mirallie E; FOThyr Group. Randomized clinical trial of ultrasonic scissors versus conventional haemostasis to compare complications and economics after total thyroidectomy (FOThyr). BJS Open. 2017 May 9;1(1):2-10. doi: 10.1002/bjs5.2. eCollection 2017 Feb. PMID 29951599